CLINICAL TRIAL: NCT07064837
Title: Conecta: A Stakeholder-informed Implementation Intervention for Contraceptive Screening, Referral, and Care Coordination.
Brief Title: Utilizing Pediatric Primary Care Connections to Advance Reproductive Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: IRB00389763; 1K23HD110615-01A1 (NIH)
Record Dates: First submitted 2025-07-07; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Contraceptive Use
Keywords: contraceptive need mothers; contraceptive need Latinas; pediatric clinic; screening; contraceptive choice; contraceptive need

STUDY DESIGN:
Intervention Model Description: One arm will be exposed to the intervention (contraceptive need screener). Other individuals will be participating in other aspects of the study (interviews, focus groups, one time survey) to help contextualize the intervention but will not receive an actual intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contraceptive need screener 'Conecta' (Experimental): The Conecta intervention is a Spanish language contraceptive need screening and referral process that includes a screener and referral to social needs navigation bundled with developmental screener in 0-12 month old pediatric well visit for written completion by the mother of the patient
  Interventions: Other: Conecta Familia; Other: Contraceptive need survey
- Historical control group (Placebo Comparator): One time survey of contraceptive use and need experience among mothers of 12-15 month olds. Recruitment will occur prior to intervention with a sample of individuals who will be comparable to those who will participate in intervention.
  Interventions: Other: Contraceptive need survey

INTERVENTIONS:
Other: Conecta Familia — The Conecta intervention is a Spanish language contraceptive need screening and referral process that includes a screener and referral to social needs navigation bundled with developmental screener in 0-12 month old pediatric well visit for written completion by the mother of the patient
  Arms: Contraceptive need screener 'Conecta'
Other: Contraceptive need survey — brief survey describing demographic information and contraceptive need, use, and experience

SUMMARY:
The purpose of this study is to understand in what ways the pediatrician's office can support women's family planning by screening for contraceptive needs at each well child visit over the first 12 months of the child's life. Part one of the study will be working with families and clinic-based social needs navigators around where and how the screening process will be integrated into an existing pediatric workflow. Part two of the study will include (a) surveying mothers of 12-15 month olds about contraceptive use experience to get a baseline followed by (b) implementing the screening process into pediatrics and measuring how well the screener is able to identify unmet contraceptive needs and how people are or are not using the screening process. This will occur over approximately 12 months. Part (b) includes enrolling families who have a contraceptive need case and following the case in the child's medical record. At the end of the 12 month intervention the investigators will (c) invite some families to participant in an interview about the experience with the contraceptive need screener. Part three will be focus group feedback from clinicians and staff about the contraceptive need screening process. Part four will be key informant interviews with community stakeholders on the expansion of this screener.

DETAILED DESCRIPTION:
The investigators propose to design and test a Spanish-language maternal contraceptive needs screening and care coordination intervention within primary care pediatrics called Conecta. The investigator's goal is to determine if this intervention can reduce unmet contraceptive need among Latina immigrant mothers. The aims of this study are:

Aim 1: To refine Conecta, a stakeholder-informed Spanish language contraceptive needs screening and care coordination intervention for implementation with existing pediatric social needs navigation, Hopkins Community Connection (HCC). The investigators will translate workflow observations into process maps and present and discuss the process maps with stakeholders who will visually assess the stakeholder's role and interaction in the workflow. Stakeholders will focus feedback on specific, practical ways that contraceptive needs screening and care coordination support would be valuable. This feedback will help the investigators build Conecta from the existing scaffolding of the HCC structure.

Aim 2: To conduct a Hybrid Type 1 implementation-effectiveness pilot of Conecta and evaluate 1) Conecta's effectiveness in reducing unmet contraceptive need, and 2) Conecta's

ELIGIBILITY:
There are four study populations categorized in this study:

* Staff of the Baltimore Medical Systems (BMS) medical practice, which includes clinicians (i.e. M.D., D.O., N.P.), medical assistants, nurses, receptionists;
* Hopkins Community Connection Resource Advocates (i.e. staff) based at the BMS;
* Community health care providers including clinicians, case managers, social workers, and nurses

Eligible BMS patients comprised of the following subpopulations:

1. Latinas with a 12 month old child who is a BMS patient;
2. Latinas with an infant 0-1 month old who is a BMS patient.

Eligibility criteria by population:

Historical control group inclusion criteria are:

* individuals who identify as Latina AND foreign-born, AND
* communication preference is Spanish AND
* 22 years or older (any parent 21 years or younger is almost always also one of the investigator's patients) AND
* are the biological parent of a 12 month old child who is a BMS patient.

Intervention cohort inclusion criteria are:

* individuals who identify as Latina AND foreign-born, AND
* communication preference is Spanish AND
* 22 years or older AND
* are the biological parent of a < 1 month old who is a BMS patient.

Participant inclusion criteria for Both:

* BMS staff OR Hopkins Community Connection Advocate staff AND
* age 18 years or older.

Participant inclusion criteria for semi-structured interviews:

* Member of intervention cohort group AND child
* has completed 12 months of life AND
* has completed contraceptive need survey.

Participant inclusion criteria for key informant interviews:

* staff member from one of 5 local health care clinics including Baltimore City Department of Health, Planned Parenthood, Women, Infants, and Children, and two federally qualified health centers AND
* direct interaction with Spanish speaking individuals AND
* age 18 years or older.

Exclusion Criteria:

Individuals with bilateral tubal ligation (permanent contraception) at time of recruitment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of unmet maternal contraceptive need | At child's 12th month of life
  Unmet need will be defined using a combination of widely used family planning and contraceptive use questions in a single survey. The same survey items will be administered to historical control group and then the cohort. There are three questions measuring contraceptive satisfaction, confidence in current contraceptive method use, and switching likelihood. These are 5 scaled answer options ranging from "very satisfied/confident to very dissatisfied/not confident at all" There are 2 possible definitions of unmet contraceptive need: 1) "Are you or your spouse or partner doing anything now to keep from getting pregnant?". 'No' and "Would you like to be using birth control right now to keep from getting pregnant? " 'Yes" and/or; 2) Low satisfaction and low confidence scores supports high likelihood of method switching and unmet need. Investigators will compare number of participants who meet unmet contraceptive need definition in cohort to number in historical control group.

SECONDARY OUTCOMES:
Feasibility of Intervention Measure (FIM) score | Baseline and 12 months of implementation
  The survey will include 4-item measures of feasibility. Score range is 4-20, higher scores indicate greater feasibility.
Acceptability of Intervention Measure (AIM) | Baseline and at 12 months of implementation
  The survey will include 4-item measures of acceptability; total mean scores range from 1 - 5, higher scores indicate greater acceptability,
Intervention Appropriateness Measure (IAM) | Baseline and at 12 months of implementation
  The survey will include 4-item measures of appropriateness. Total mean scores 1-5, higher score indicates greater appropriateness,
Number of clinic staff engaged with the intervention | Up to 15 months post intervention
  As part of implementation evaluation investigators will conduct a focus group using the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) framework.

CONTACTS AND LOCATIONS:
Overall Officials: Tania Caballero, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Baltimore Medical Systems Yard 56, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No